CLINICAL TRIAL: NCT06283810
Title: The Effects of Interpersonal Relationship Psychotherapy and Laughter Therapy on Interpersonal Relationships, Problem Solving and Self-Reflection in Midwifery Students
Brief Title: The Effects of Interpersonal Relationship Psychotherapy and Laughter Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/168
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Midwifery Students
Keywords: self reflection; interpersonel relationship; laughter therapy
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- psychotherapy of interpersonal relationships (Experimental): "Informed Consent Form" and "Voluntary Consent Form" will be presented to the students assigned to Group 1 in the first interview and their consent will be obtained, "Student Information Form (ANNEX-1)", "CIBS (ANNEX-3)", PCI (ANNEX-4), CPI (ANNEX-5) and SB3S (ANNEX-6) will be applied.
  After the initial data are collected, 2-3 sessions of individual interviews will be conducted to assess the student's suitability for Group CIPT.
  Interventions: Behavioral: psychotherapy of interpersonal relationships
- laughter therapy (Experimental): In the first interview, "Informed Consent Form" and "Voluntary Consent Form" will be presented to the students assigned to Group 2 and their consent will be obtained, and "Student Information Form (ANNEX-1)", "CIBS (ANNEX-3)", PCI (ANNEX-4), CPI (ANNEX-5) and SB3S (ANNEX-6) will be applied.
  After the initial data were collected, the students in Experiment 2 will be informed about Laughter Therapy and Group IPT. An agreement will be made with the students about the points to be considered regarding laughter therapy
  Interventions: Behavioral: laughter therapy
- Plasebo group (Placebo Comparator): "Informed Consent Form" and "Voluntary Consent Form" were presented to the students in the placebo group in the first interview and their consent was obtained, "Student Information Form (ANNEX-1)", "CIBS (ANNEX-3)", PCI (ANNEX-4), CPI (ANNEX-5) and SB3S (ANNEX-6) were applied.
  Interventions: Behavioral: Plasebo
- control group (No Intervention): The students assigned to G4 will be informed that they are in the control group and that no application will be made. After the completion of the study data (by giving information about Group CIPT and laughter therapy), it will be stated that they can receive Group CIPT or laughter therapy if they wish.

INTERVENTIONS:
Behavioral: psychotherapy of interpersonal relationships — Group KIPT will be 1 session per week and each session will last 90 minutes. There will be 7 sessions in total, and a completion session will be held 2 weeks after the completion of Group KIPT. In order for the students in G1 to understand which group they are in, they will also be informed about the points to be considered regarding laughter therapy. An unstructured laughter intervention will be applied at the beginning or at the end of the sessions in which group IPT is applied.
  Measurements will be made using "ANNEX-3, ANNEX-4, ANNEX-5, ANNEX-6" in the 4th week (intervention interval), 8th week (end of intervention) and 12th week (long-term effect). Within the scope of work packages 3 and 4, KIPT application and other measurements will be made.
  Arms: psychotherapy of interpersonal relationships
Behavioral: laughter therapy — Laughter therapy is 1 session per week and each session will last 40 minutes. A total of 8 sessions will continue. Each session will start with warm-up and deep breathing exercises and will continue with applause and childish games. Afterwards, games specific to each session will be added. Unstructured interviews will be conducted with G2 at the beginning or at the end of the session, suggesting that they were subjected to group CIPT. Measurements will be made using "ANNEX-3, ANNEX-4, ANNEX-5, ANNEX-6" in the 4th week (intervention interval), 8th week (end of intervention) and 12th week (long-term effect) when the interviews start.
  Arms: laughter therapy
Behavioral: Plasebo — After the initial data are collected, unstructured interviews about the interpersonal relationships of the person will be conducted by conducting individual interviews with each student for 2-3 sessions at the beginning of the study in case the student does not understand which group he/she is in. Afterwards, unstructured random interviews and laughter intervention will be conducted for a total of 8 sessions lasting 40 minutes, 1 session per week. Measurements will be made using "ANNEX-3, ANNEX-4, ANNEX-5, ANNEX-6" in the 4th week, 8th week and 12th week (long-term effect) when the interviews start.
  Arms: Plasebo group

SUMMARY:
Midwives, who have an important place in the health system, are expected to be equipped to meet the health care needs of women (Fışkın & Doğan, 2020). Therefore, midwifery students, who are known to play a role in promoting women's health, should have good interpersonal relationships, good problem-solving skills, and high self-reflection and insight, which are assumed to be effective in both, in order to fulfill these responsibilities.

Translated with DeepL.com (free version)

DETAILED DESCRIPTION:
Self-reflection supports the development of strategies for self-monitoring and professional competence by improving problem-solving skills. Self-reflection serves as an important building block in the integration and structuring of experience and sense of self, as well as providing continuity, coherence and meaning to life. It is thought that midwives with self-reflection will be more logical, healthy, happy and successful. It is seen that midwives with high self-reflection are dedicated to lifelong learning, examining, reflecting and developing, and develop personally and professionally (Bass et al., 2022). The quality of care will increase as midwives who develop self-reflection can observe, investigate, evaluate and discover events with a realistic eye while providing care, thus the midwifery profession will progress as a scientific discipline.

ELIGIBILITY:
Inclusion Criteria:

* - To be a 1st, 2nd and 3rd year student of Istanbul University-Cerrahpaşa Faculty of Health Sciences, Department of Midwifery.
* To get less than 2 points from the "General Health Questionnaire".

Exclusion Criteria:

* - Those with an indifferent attachment style,
* Those with antisocial or narcissistic traits,
* Those with active suicidal thoughts,
* People with psychiatric diagnosis and medication,
* Those with urinary incontinence,
* Those with severe back pain,
* Those who have undergone surgical operation within the last 1 year.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
self-reflection skills | 12 week
  It is thought that self-reflection plays a mediating role in the interpersonal relationships and problem solving skills of the students in the study. For this reason, it was decided to determine the self-reflection characteristics of the students, but a suitable scale could not be found. Thus, it was decided to develop a scale to determine the self-reflection characteristics of students studying in Health Sciences. In this direction, the scale development study was carried out by obtaining the approval of Istanbul University-Cerrahpaşa Social and Human Sciences Research Ethics Committee (2023/120) and the necessary permission from Istanbul University-Cerrahpaşa Faculty of Health Sciences Dean's Office (06.10.2023-802307).
problem solving skills | 12 week
  Problem Solving Inventory was developed by Heppner and Peterson (1982). It was adapted into Turkish by Taylan (1990), Şahin, Şahin and Heppner (1993). The scale is a six-point Likert-type scale consisting of 35 items and three factors. The first of the three factors is problem solving confidence (11 items), the second is problem avoidance/approach (16 items), and the third is control (15 items). Scale options are scored between one and six as "I always behave like this" and "I never behave like this".
interpersonal relationship skills | 12 week
  Interpersonal Relationship Dimension Scale (IRDS; ANNEX-3): This scale was developed by İmamoğlu and Aydın (2009). The IBS is a 5-point Likert-type scale consisting of 53 items, which is suitable for Turkish conditions, analyses interpersonal relationships and determines relationship dimensions. The scale consists of four sub-dimensions: Consent Dependence, Empathy, Trust in Others and Emotion Awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Namazinia M, Mazlum SR, Mohajer S, Lopez V. Effects of laughter yoga on health-related quality of life in cancer patients undergoing chemotherapy: a randomized clinical trial. BMC Complement Med Ther. 2023 Jun 12;23(1):192. doi: 10.1186/s12906-023-04028-2. PMID 37303065